CLINICAL TRIAL: NCT00454259
Title: Fentanyl Ultra Low Doses Effects on Human Volunteer's Nociceptive Threshold. Towards a Simple Pharmacological Test Able to Predict Pain Vulnerability, Post Operative Hyperalgesia Development Risk?
Brief Title: Fentanyl Ultra Low Doses Effects on the Nociceptive Threshold
Acronym: FENTANULD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Jean-Pierre LEROY / Clinical Research and Innovation Director, University Hospital, Bordeaux
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: CHUBX 2006/08
Record Dates: First submitted 2007-03-29; First posted 2007-03-30 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2007-03

CONDITIONS: Pain, Postoperative
Keywords: Postoperative Hyperalgesia; Human volunteer; Fentanyl; Randomized Controlled Trial; Pain chronicisation; Predictive test
MeSH Terms: conditions — Pain, Postoperative | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): 0,5 µg/kg
  Interventions: Drug: Fentanyl/Placebo injection
- 2 (Experimental): 0,05 µg/kg
  Interventions: Drug: Fentanyl/Placebo injection
- 3 (Experimental): 0,005 µg/kg
  Interventions: Drug: Fentanyl/Placebo injection
- 4 (Placebo Comparator): NaCl 0,9 %
  Interventions: Drug: Fentanyl/Placebo injection

INTERVENTIONS:
Drug: Fentanyl/Placebo injection — Ultra low dose intravenous injection

SUMMARY:
Exaggerated pain and hyperalgesia are major issues after surgery and can lead to chronic pain. Opioid are parts of pain sensitization processes but remain absolutely necessary in the intraoperative period. NMDA receptor antagonists succeed in reducing this pain sensitization process. Recent studies show that in pain and opioid-experienced rats (POER) fentanyl ultra low doses do not induce analgesia, as observed in naive rats, but hyperalgesia. This is the first demonstration that a drug can induce opposite effect depending on individual history. We also observed a strong correlation between this hyperalgesic response in POER and the intensity of hyperalgesia they develop later, after inflammatory or surgical pain. The main aim of this study is to measure the dose effect response to fentanyl "ultra low doses" on human volunteer's nociceptive threshold, to determine if such an opposite response profile can be revealed.

DETAILED DESCRIPTION:
* Principal Objective : "Evaluate fentanyl "ultra low doses" effects on human volunteer's nociceptive threshold depending on their prior pain and opioid experience."
* Secondary Objective : "Confirm the innocuousness of this test (the 3 "ultra low doses" used in this trial will be 10 to 1,000 fold lower than low doses use for anesthesia and analgesia) and to find the fentanyl ultra low dose that could be used to develop a pain sensitisation predictive test."
* Study design : Bicentric, prospective, randomized, double-blind study.

Inclusion criteria :

In both groups:

* 18-40 years old male volunteer
* weight: 60 to 85 kg
* ASA score: 1
* Informed consent obtained from the patient
* Gender : Male

In "operated" group:

- At least one history of peripheral surgery under general anesthesia with opioid in the past five years

Exclusion criteria :

In both groups:

* The patient do not accept inclusion to the study
* Drug or alcohol abuse history
* Chronic use of analgesic drugs or history of chronic pain
* Analgesic or opioid consumption within the 12hs preceding the fentanyl or placebo injection
* Neurological and/or psychiatric disorder, inability to give informed consent
* Psychological trauma within the two year preceding the inclusion
* Any contraindication to fentanyl use
* Use of any medication interacting with fentanyl
* Exclusion period from the national healthy volunteer register
* Gender : Female

In "healthy" group:

- Any history of general anesthesia or surgery

* Study plan: comparing two groups that only defer by their surgical and opioid prior experience and will receive three fentanyl ultra low doses (10 to 1,000 fold lower than low doses use for anesthesia and analgesia) and placebo (cross over administration, one week wash out period).
* Number of subjects : 48

ELIGIBILITY:
Inclusion Criteria:

In both groups:

* 18-40 years old male volunteer
* Weight: 60 to 85 kg
* ASA score: 1
* Informed consent obtained from the patient

In "operated" group:

* At least one history of peripheral surgery under general anesthesia with opioid in the past five years.

Exclusion Criteria:

In both groups:

* The patients do not accept inclusion to the study
* Drug or alcohol abuse history
* Chronic use of analgesic drugs or history of chronic pain
* Analgesic or opioid consumption within the 12hs preceding the fentanyl or placebo injection
* Neurological and/or psychiatric disorder, inability to give informed consent
* Psychological trauma within the two year preceding the inclusion
* Any contraindication to fentanyl use
* Use of any medication interacting with fentanyl
* Exclusion period from the national healthy volunteer register

In "healthy" group:

* Any history of general anesthesia or surgery

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2007-03; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Nociceptive threshold evaluated with sternal electronical Von Frey mechanical stimulation. The stimulation will increase until the volunteer presses a trigger when the stimulation becomes painful. | 5 min after injection, and every 15 min during 1 hour

SECONDARY OUTCOMES:
Non invasive blood pressure (SBP, DBP), heart rate, respiratory rate, pulse oxymetry and cognitive functions evaluation (sedation score). | all along the experimentation

CONTACTS AND LOCATIONS:
Overall Officials: Philippe RICHEBE, Dr, Study Director — University Hospital, Bordeaux; Gérard JANVIER, PHD, Principal Investigator — University Hospital, Bordeaux; Claude DUBRAY, PHD, Principal Investigator — University Hospital, Bordeaux; Alain ESCHALIER, PHD, Principal Investigator — University Hospital, Bordeaux; jean DUALE CHRISTIAN, Dr, Principal Investigator — University Hospital, Bordeaux; Gisèle PICKERING, Dr, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux Département d'Anesthésie-Réanimation II, Pessac, Hôpital Cardiologique, France

REFERENCES:
- [Background] Hsu YW, Somma J, Hung YC, Tsai PS, Yang CH, Chen CC. Predicting postoperative pain by preoperative pressure pain assessment. Anesthesiology. 2005 Sep;103(3):613-8. doi: 10.1097/00000542-200509000-00026. PMID 16129988
- [Background] Kalkman JC, Visser K, Moen J, Bonsel JG, Grobbee ED, Moons MKG. Preoperative prediction of severe postoperative pain. Pain. 2003 Oct;105(3):415-423. doi: 10.1016/S0304-3959(03)00252-5. PMID 14527702
- [Background] Perkins FM, Kehlet H. Chronic pain as an outcome of surgery. A review of predictive factors. Anesthesiology. 2000 Oct;93(4):1123-33. doi: 10.1097/00000542-200010000-00038. No abstract available. PMID 11020770
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] Celerier E, Laulin JP, Corcuff JB, Le Moal M, Simonnet G. Progressive enhancement of delayed hyperalgesia induced by repeated heroin administration: a sensitization process. J Neurosci. 2001 Jun 1;21(11):4074-80. doi: 10.1523/JNEUROSCI.21-11-04074.2001. PMID 11356895
- [Background] Coderre TJ, Katz J, Vaccarino AL, Melzack R. Contribution of central neuroplasticity to pathological pain: review of clinical and experimental evidence. Pain. 1993 Mar;52(3):259-285. doi: 10.1016/0304-3959(93)90161-H. PMID 7681556
- [Background] Shen KF, Crain SM. Cholera toxin-B subunit blocks excitatory effects of opioids on sensory neuron action potentials indicating that GM1 ganglioside may regulate Gs-linked opioid receptor functions. Brain Res. 1990 Oct 29;531(1-2):1-7. doi: 10.1016/0006-8993(90)90751-v. PMID 1981160
- [Background] Crain SM, Shen KF. Modulation of opioid analgesia, tolerance and dependence by Gs-coupled, GM1 ganglioside-regulated opioid receptor functions. Trends Pharmacol Sci. 1998 Sep;19(9):358-65. doi: 10.1016/s0165-6147(98)01241-3. PMID 9786023
- [Background] Richebe P, Rivat C, Laulin JP, Maurette P, Simonnet G. Ketamine improves the management of exaggerated postoperative pain observed in perioperative fentanyl-treated rats. Anesthesiology. 2005 Feb;102(2):421-8. doi: 10.1097/00000542-200502000-00028. PMID 15681961
- [Background] Woolf CJ, Salter MW. Neuronal plasticity: increasing the gain in pain. Science. 2000 Jun 9;288(5472):1765-9. doi: 10.1126/science.288.5472.1765. PMID 10846153
- [Background] Rivat C, Laulin JP, Corcuff JB, Celerier E, Pain L, Simonnet G. Fentanyl enhancement of carrageenan-induced long-lasting hyperalgesia in rats: prevention by the N-methyl-D-aspartate receptor antagonist ketamine. Anesthesiology. 2002 Feb;96(2):381-91. doi: 10.1097/00000542-200202000-00025. PMID 11818772
- [Background] Simonnet G, Rivat C. Opioid-induced hyperalgesia: abnormal or normal pain? Neuroreport. 2003 Jan 20;14(1):1-7. doi: 10.1097/00001756-200301200-00001. No abstract available. PMID 12544821